CLINICAL TRIAL: NCT01119625
Title: Evaluation of Immunological Persistence Following 3-dose Priming With GSK Biologicals' 10-valent Pneumococcal Conjugate Vaccine in Study NCT00808444 and Safety and Immunogenicity Following a Booster Dose of the Same Vaccine
Brief Title: Immunological Persistence After Priming With GSK1024850A Vaccine and Safety& Immunogenicity After Booster Dose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113266
Record Dates: First submitted 2010-04-22; First posted 2010-05-07 (Estimated); Results first posted 2012-03-22 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2016-09

CONDITIONS: Infections, Streptococcal
Keywords: safety; Streptococcus pneumoniae; immunogenicity; Pneumococcal conjugate vaccine; Haemophilus influenzae
MeSH Terms: conditions — Streptococcal Infections; Haemophilus Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (2):
- Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group (Experimental): children primed with 3 doses of commercial lot of Synflorix™ co-administered with Rotarix™ and Infanrix™-hexa in the primary phase of the study (NCT00808444) and boosted with commercial lot of Synflorix™ co-administered with Infanrix™-IPV/Hib. The Synflorix™ vaccine (commercial lots) was administered intramuscularly in the right deltoid or anterolateral thigh and the Infanrix™-IPV/Hib vaccine was administered intramuscularly in the left deltoid or anterolateral thigh.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A; Biological: Infanrix-IPV/Hib
- Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group (Active Comparator): children primed with 3 doses of clinical lot of Synflorix™ + Rotarix™ co-administered with Infanrix™-hexa in the primary phase of the study (NCT00808444) and boosted with commercial lot of Synflorix™ co-administered with Infanrix™-IPV/Hib. The Synflorix™ vaccine (clinical and commercial lots) was administered intramuscularly in the right deltoid or anterolateral thigh and the Infanrix™-IPV/Hib vaccine was administered intramuscularly in the left deltoid or anterolateral thigh.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A; Biological: Infanrix-IPV/Hib

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK1024850A — Intramuscular injection, one dose
Biological: Infanrix-IPV/Hib — Intramuscular injection, one dose

SUMMARY:
This primary purpose of this study is the evaluation of the immunological persistence following completion of the 3-dose primary vaccination course with either a clinical or a commercial lot of pneumococcal conjugate vaccine GSK1024850A in study NCT00808444. In addition, the study will also assess the safety, reactogenicity and immunogenicity of a fourth dose of pneumococcal conjugate vaccine GSK1024850A (commercial lot) when co-administered with Infanrix-IPV/Hib at 18-21 months of age in children primed in study NCT00808444.

The primary vaccination study was conducted in Malaysia and Singapore. The booster vaccination study will not be performed in Malaysia since the pneumococcal conjugate vaccine GSK1024850A has been registered in September 2009. However, subjects in Malaysia will be offered a booster dose of the commercial pneumococcal conjugate vaccine licensed in Malaysia and Infanrix-IPV/Hib vaccine during the second year of life according to the nationally recommended regimen. Administration of the booster dose will be outside the set-up of a clinical trial. Hence no data will be collected, no blood samples will be taken in Malaysia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol
* Male or female between, and including, 18 and 21 months of age at the time of booster vaccination.
* Subjects who received three doses of pneumococcal conjugate vaccine in study NCT00808444
* Written informed consent obtained from the parents/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding vaccination, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to vaccination.
* A family history of congenital or hereditary immunodeficiency.
* Administration of immunoglobulins and/ or any blood products within the 3 months preceding vaccination or planned use during the study period.
* Administration of any pneumococcal and/or vaccine containing diphtheria, tetanus, pertussis, poliomyelitis or Haemophilus influenzae type b antigens since the end of study NCT00808444.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the study period starting from 30 days before vaccination and ending 30 days after vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of any reaction or allergic disease likely to be exacerbated by any component of the study vaccines.
* Known hypersensitivity to any component of the study vaccines including anaphylactic reactions following the administration of the study vaccines.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures. (Subjects who have had a single uncomplicated febrile convulsion in the past can be included)
* Fever at the time of vaccination.

  * Fever is defined as rectal temperature >= 38.0°C or tympanic/axillary/ oral temperature >= 37.5°C.
* Acute disease at the time of enrolment.

  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Child in care.

Ages: 18 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 238 (Actual)
Dates: Start 2010-07-12; Primary Completion 2011-02-17 (Actual); Study Completion 2011-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lim FS, Koh MT, Tan KK, Chan PC, Chong CY, Shung Yehudi YW, Teoh YL, Shafi F, Hezareh M, Swinnen K, Borys D. A randomised trial to evaluate the immunogenicity, reactogenicity, and safety of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) co-administered with routine childhood vaccines in Singapore and Malaysia. BMC Infect Dis. 2014 Oct 2;14:530. doi: 10.1186/1471-2334-14-530. PMID 25278086
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This booster study was conducted in Singapore only wheras the primary vaccination phase (NCT00808444) was conducted in Singapore and Malaysia.
Groups:
- Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group: children primed with 3 doses of commercial lot of Synflorix™ co-administered with Rotarix™ and Infanrix™-hexa in the primary phase of the study (NCT00808444) and boosted with commercial lot of Synflorix™ co-administered with Infanrix™-IPV/Hib. The Synflorix™ vaccine (clinical and commercial lots) was administered intramuscularly in the right deltoid or anterolateral thigh and the Infanrix™-IPV/Hib vaccine was administered intramuscularly in the left deltoid or anterolateral thigh.
Period: Overall Study
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Started | 118 | 120
Completed | 115 | 116
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group | Total
Number analyzed (Participants) | 118 | 120 | 238
Age, Continuous [Mean (Standard Deviation); unit: Months] | 18.8 (0.84) | 18.9 (0.87) | 18.9 (0.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 49 | 111
  Male | 56 | 71 | 127

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes.
Description: Vaccine pneumococcal serotypes assessed were serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
  Concentrations were expressed as geometric mean concentrations (GMCs) in microgram per millilitre (µg/mL).
  Pneumococcal serotype specific total imunoglobuline G (IgG) antibodies were measured by 22F-inhibition Enzyme-linked immunosorbent assay (ELISA). The cut-off of the assay was 0.05 µg/mL.
Time Frame: Before booster vaccination at Month 0
Population: The analysis was performed on the According-To-Protocol cohort for analysis of antibody persistence which included subjects primed in the primary study (NCT00808444) and for whom assay results were available for antibodies against at least 1 vaccine antigen component for the blood sampling taken before the administration of the booster dose.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 111 | 112
µg/mL
  Anti-1 [Pre-booster] | 0.48 [0.40 to 0.57] | 0.35 [0.30 to 0.41]
  Anti-4 [Pre-booster]: number analyzed (Participants) | 107 | 106
  Anti-4 [Pre-booster] | 0.56 [0.48 to 0.67] | 0.48 [0.40 to 0.58]
  Anti-5 [Pre-booster]: number analyzed (Participants) | 103 | 103
  Anti-5 [Pre-booster] | 0.76 [0.65 to 0.89] | 0.54 [0.47 to 0.63]
  Anti-6B [Pre-booster]: number analyzed (Participants) | 103 | 102
  Anti-6B [Pre-booster] | 0.34 [0.29 to 0.40] | 0.32 [0.25 to 0.41]
  Anti-7F [Pre-booster]: number analyzed (Participants) | 104 | 105
  Anti-7F [Pre-booster] | 0.88 [0.75 to 1.03] | 0.91 [0.78 to 1.07]
  Anti-9V [Pre-booster]: number analyzed (Participants) | 105 | 102
  Anti-9V [Pre-booster] | 0.90 [0.77 to 1.06] | 0.73 [0.62 to 0.85]
  Anti-14 [Pre-booster]: number analyzed (Participants) | 105 | 100
  Anti-14 [Pre-booster] | 1.06 [0.86 to 1.31] | 0.91 [0.75 to 1.11]
  Anti-18C [Pre-booster]: number analyzed (Participants) | 109 | 108
  Anti-18C [Pre-booster] | 0.83 [0.69 to 1.01] | 0.78 [0.65 to 0.93]
  Anti-19F [Pre-booster]: number analyzed (Participants) | 103 | 103
  Anti-19F [Pre-booster] | 1.10 [0.87 to 1.40] | 0.96 [0.82 to 1.13]
  Anti-23F [Pre-booster]: number analyzed (Participants) | 108 | 106
  Anti-23F [Pre-booster] | 0.66 [0.51 to 0.84] | 0.47 [0.38 to 0.58]

2. Primary Outcome: Concentrations of Antibodies Against Protein D (PD).
Description: Anti-PD antibodies were determined using an ELISA assay. Concentration of specific PD antibodies was determined, using a standard reference serum. The cut-off of the assay is 100 ELISA units per millilitre (EU/mL).
Time Frame: Before booster vaccination at Month 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 116 | 118
EU/mL | 801.6 [693.1 to 927.1] | 619.7 [530.1 to 724.3]

3. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs).
Description: Solicited AEs = AEs to be recorded as endpoints in the clinical study. The presence/occurrence/intensity of these events is actively solicited from the subject or an observer during a specified post-vaccination follow-up period.
  Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling above 30 millimetre (mm).
Time Frame: Within 4 days (Days 0-3) after booster vaccination.
Population: The analysis of safety was performed on the Total vaccinated cohort which included all subjects with booster dose administration documented. The analysis of the solicited symptoms based on the Total Vaccinated cohort included subjects with documented safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 117 | 117
Participants
  Any pain | 61 | 70
  Grade 3 pain | 8 | 13
  Any redness | 66 | 61
  Grade 3 redness | 0 | 0
  Any swelling | 45 | 49
  Grade 3 swelling | 1 | 0

4. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Adverse Events (AEs).
Description: Solicited general symptoms assessed were drowsiness, irritability, loss of appetite and fever (= axillary temperature equal to or above 37.5 degrees Celsius (°C)).
  Any= occurrence of any general symptom regardless of intensity grade or relationship to vaccination Grade 3 drowsiness = drowsiness which prevented normal activity. Grade 3 irritability = crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 fever = temperature >39.5°C.
  Related = solicited symptom assessed by the investigator as causally related to study vaccination.
Time Frame: Within 4 days (Days 0-3) after booster vaccination.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 117 | 117
Participants
  Any drowsiness | 38 | 49
  Grade 3 drowsiness | 2 | 2
  Related drowsiness | 38 | 48
  Fever >= 37.5°C | 56 | 75
  Fever > 39.5°C | 1 | 1
  Related fever | 55 | 72
  Any irritability | 51 | 67
  Grade 3 irritability | 3 | 5
  Related irritability | 50 | 67
  Any loss of appetite | 42 | 49
  Grade 3 loss of appetite | 1 | 1
  Related loss of appetite | 41 | 47

5. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs).
Description: Unsolicited AEs = Any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: Within 31 days (Days 0-30) after booster vaccination
Population: The analysis of safety was performed on the Total vaccinated cohort which included all subjects with booster dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 118 | 120
Participants | 18 | 25

6. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: During the entire study period, from the booster vaccination, at Month 0, up to the study end, at Month 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 118 | 120
Participants | 0 | 4

7. Secondary Outcome: Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes.
Description: Opsonophagocytic activity (OPA) testing was not performed.
Time Frame: Before and one month after booster vaccination (at Month 0 and Month 1)
Reporting Status: Not Posted, anticipated posting 2099-12

8. Secondary Outcome: Opsonophagocytic Activity Against Cross-reactive Pneumococcal Serotypes 6A and 19A.
Description: Opsonophagocytic activity (OPA) testing was not performed.
Time Frame: Before and one month after booster vaccination (at Month 0 and Month 1)
Reporting Status: Not Posted, anticipated posting 2099-12

9. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes.
Description: Cross-reactive pneumococcal serotypes assessed were serotypes 6A and 19A. Concentrations were expressed as geometric mean concentrations (GMCs) in microgram per millilitre (µg/mL).
  The antibody concentrations against the cross-reactive pneumococcal serotypes 6A and 19A were determined by 22F-inhibition Enzyme-linked immunosorbent assay (ELISA). The cut-off of the assay was 0.05 µg/mL.
Time Frame: Before booster vaccination at Month 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 112 | 111
µg/mL
  Anti-6A [pre-booster]: number analyzed (Participants) | 109 | 111
  Anti-6A [pre-booster] | 0.23 [0.18 to 0.28] | 0.21 [0.16 to 0.26]
  Anti-19A [pre-booster]: number analyzed (Participants) | 112 | 109
  Anti-19A [pre-booster] | 0.18 [0.14 to 0.22] | 0.19 [0.15 to 0.24]

10. Secondary Outcome: Concentrations of Antibodies Against Diphtheria and Tetanus.
Description: Concentrations were expressed as geometric mean concentrations (GMCs) in International units per millilitre (IU/mL). The cut-off of the assay was 0.1 IU/mL.
Time Frame: Before booster vaccination at Month 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 43 | 49
IU/mL
  Anti-diphtheria [pre-booster]: number analyzed (Participants) | 42 | 49
  Anti-diphtheria [pre-booster] | 0.32 [0.25 to 0.39] | 0.30 [0.24 to 0.39]
  Anti-tetanus [pre-booster]: number analyzed (Participants) | 43 | 48
  Anti-tetanus [pre-booster] | 0.51 [0.43 to 0.61] | 0.47 [0.38 to 0.59]

11. Secondary Outcome: Concentrations of Antibodies Against Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN).
Description: Concentrations were expressed as geometric mean concentrations (GMCs) in ELISA units per millilitre (EU/mL). The cut-off of the assay was 5 EU/mL.
Time Frame: Before booster vaccination at Month 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 42 | 47
EU/mL
  Anti-PT [pre-booster]: number analyzed (Participants) | 41 | 45
  Anti-PT [pre-booster] | 5.7 [4.5 to 7.2] | 6.5 [4.7 to 8.9]
  Anti-FHA [pre-booster]: number analyzed (Participants) | 40 | 46
  Anti-FHA [pre-booster] | 19.5 [15.1 to 25.3] | 29.2 [21.5 to 39.6]
  Anti-PRN [pre-booster] | 14.8 [10.7 to 20.6] | 15.1 [11.1 to 20.5]

12. Secondary Outcome: Concentrations of Antibodies Against Polyribosyl-ribitol Phosphate (PRP).
Description: Concentrations were expressed as geometric mean concentrations (GMCs) in microgram per millilitre (µg/mL). The cut-off of the assay was 0.15 µg/mL.
Time Frame: Before booster vaccination at Month 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 52 | 57
µg/mL | 0.68 [0.50 to 0.92] | 0.85 [0.65 to 1.11]

13. Secondary Outcome: Titers of Antibodies Against Poliovirus Types 1, 2 and 3.
Description: Titers were expresses as geometric mean titers (GMTs). The cut-off of the assay was 8.
Time Frame: Before booster vaccination at Month 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 29 | 25
Titers
  Anti-polio 1 [pre-booster] | 40.7 [23.2 to 71.3] | 32.8 [19.1 to 56.3]
  Anti-polio 2 [pre-booster] | 38.7 [26.5 to 56.7] | 34.9 [18.8 to 64.7]
  Anti-polio 3 [pre-booster] | 40.7 [24.4 to 67.8] | 43.3 [24.0 to 78.0]

14. Secondary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes.
Description: as for outcome 1
Time Frame: Before and one month after booster vaccination (at Month 0 and Month 1)
Population: The ATP cohort for immunogenicity included evaluable subjects for whom assay results were available for antibodies against at least 1 study vaccine antigen component after booster vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 109 | 111
µg/mL
  Anti-1 [pre-booster]: number analyzed (Participants) | 109 | 109
  Anti-1 [pre-booster] | 0.48 [0.40 to 0.57] | 0.35 [0.30 to 0.41]
  Anti-1 [post-booster]: number analyzed (Participants) | 107 | 111
  Anti-1 [post-booster] | 7.14 [6.12 to 8.32] | 6.29 [5.38 to 7.35]
  Anti-4 [pre-booster]: number analyzed (Participants) | 105 | 103
  Anti-4 [pre-booster] | 0.56 [0.47 to 0.67] | 0.48 [0.40 to 0.58]
  Anti-4 [post-booster]: number analyzed (Participants) | 106 | 109
  Anti-4 [post-booster] | 7.53 [6.44 to 8.80] | 7.43 [6.33 to 8.71]
  Anti-5 [pre-booster]: number analyzed (Participants) | 101 | 100
  Anti-5 [pre-booster] | 0.77 [0.65 to 0.90] | 0.54 [0.46 to 0.62]
  Anti-5 [post-booster]: number analyzed (Participants) | 106 | 108
  Anti-5 [post-booster] | 7.91 [6.91 to 9.06] | 7.16 [6.25 to 8.20]
  Anti-6B [pre-booster]: number analyzed (Participants) | 101 | 99
  Anti-6B [pre-booster] | 0.34 [0.29 to 0.40] | 0.32 [0.25 to 0.41]
  Anti-6B [post-booster]: number analyzed (Participants) | 106 | 109
  Anti-6B [post-booster] | 3.30 [2.85 to 3.81] | 3.12 [2.59 to 3.76]
  Anti-7F [pre-booster]: number analyzed (Participants) | 102 | 102
  Anti-7F [pre-booster] | 0.88 [0.75 to 1.04] | 0.93 [0.80 to 1.08]
  Anti-7F [post-booster]: number analyzed (Participants) | 106 | 109
  Anti-7F [post-booster] | 9.02 [7.77 to 10.47] | 9.25 [8.04 to 10.64]
  Anti-9V [pre-booster]: number analyzed (Participants) | 103 | 99
  Anti-9V [pre-booster] | 0.90 [0.77 to 1.06] | 0.72 [0.62 to 0.84]
  Anti-9V [post-booster]: number analyzed (Participants) | 107 | 109
  Anti-9V [post-booster] | 9.36 [8.15 to 10.75] | 10.42 [8.94 to 12.14]
  Anti-14 [pre-booster]: number analyzed (Participants) | 103 | 97
  Anti-14 [pre-booster] | 1.05 [0.85 to 1.31] | 0.93 [0.76 to 1.14]
  Anti-14 [post-booster]: number analyzed (Participants) | 106 | 106
  Anti-14 [post-booster] | 13.03 [10.95 to 15.50] | 13.28 [11.06 to 15.95]
  Anti-18C [pre-booster]: number analyzed (Participants) | 107 | 105
  Anti-18C [pre-booster] | 0.83 [0.69 to 1.01] | 0.78 [0.66 to 0.94]
  Anti-18C [post-booster]: number analyzed (Participants) | 106 | 108
  Anti-18C [post-booster] | 19.80 [17.02 to 23.03] | 24.19 [20.66 to 28.33]
  Anti-19F [pre-booster]: number analyzed (Participants) | 101 | 100
  Anti-19F [pre-booster] | 1.11 [0.87 to 1.41] | 0.97 [0.82 to 1.14]
  Anti-19F [post-booster]: number analyzed (Participants) | 106 | 108
  Anti-19F [post-booster] | 19.68 [17.22 to 22.51] | 20.55 [17.62 to 23.98]
  Anti-23F [pre-booster]: number analyzed (Participants) | 106 | 103
  Anti-23F [pre-booster] | 0.65 [0.50 to 0.83] | 0.47 [0.38 to 0.59]
  Anti-23F [post-booster]: number analyzed (Participants) | 107 | 109
  Anti-23F [post-booster] | 7.19 [5.94 to 8.71] | 6.83 [5.77 to 8.07]

15. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes.
Description: as for outcome 9
Time Frame: Before and one month after booster vaccination (at Month 0 and Month 1)
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 110 | 109
µg/mL
  Anti-6A [pre-booster]: number analyzed (Participants) | 107 | 108
  Anti-6A [pre-booster] | 0.23 [0.18 to 0.28] | 0.21 [0.16 to 0.26]
  Anti-6A [post-booster]: number analyzed (Participants) | 106 | 108
  Anti-6A [post-booster] | 2.13 [1.70 to 2.66] | 1.99 [1.60 to 2.49]
  Anti-19A [pre-booster]: number analyzed (Participants) | 110 | 106
  Anti-19A [pre-booster] | 0.18 [0.14 to 0.22] | 0.20 [0.15 to 0.25]
  Anti-19A [post-booster]: number analyzed (Participants) | 106 | 109
  Anti-19A [post-booster] | 2.13 [1.65 to 2.76] | 2.96 [2.26 to 3.87]

16. Secondary Outcome: Concentrations of Antibodies Against Protein D (PD).
Description: as for outcome 2
Time Frame: Before and one month after booster vaccination (at Month 0 and Month 1)
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 113 | 115
EU/mL
  Anti-PD [pre-booster] | 794.9 [686.3 to 920.7] | 618.4 [527.8 to 724.6]
  Anti-PD [post-booster]: number analyzed (Participants) | 107 | 111
  Anti-PD [post-booster] | 3631.3 [3149.2 to 4187.2] | 3115.9 [2634.7 to 3685.1]

17. Secondary Outcome: Concentrations of Antibodies Against Diphtheria and Tetanus.
Description: as for outcome 10
Time Frame: Before and one month after booster vaccination (at Month 0 and Month 1)
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 52 | 55
IU/mL
  Anti-diphtheria [pre-booster]: number analyzed (Participants) | 41 | 47
  Anti-diphtheria [pre-booster] | 0.31 [0.25 to 0.39] | 0.29 [0.23 to 0.37]
  Anti-diphtheria [post-booster] | 8.17 [6.72 to 9.94] | 10.89 [9.16 to 12.94]
  Anti-tetanus [pre-booster]: number analyzed (Participants) | 42 | 46
  Anti-tetanus [pre-booster] | 0.52 [0.43 to 0.62] | 0.46 [0.37 to 0.58]
  Anti-tetanus [post-booster] | 14.35 [12.41 to 16.60] | 14.73 [12.75 to 17.01]

18. Secondary Outcome: Concentrations of Antibodies Against Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN).
Description: as for outcome 11
Time Frame: Before and one month after booster vaccination (at Month 0 and Month 1)
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 52 | 55
EU/mL
  Anti-PT [pre-booster]: number analyzed (Participants) | 40 | 43
  Anti-PT [pre-booster] | 5.8 [4.5 to 7.3] | 6.8 [4.9 to 9.3]
  Anti-PT [post-booster] | 80.8 [65.6 to 99.4] | 86.0 [67.9 to 108.9]
  Anti-FHA [pre-booster]: number analyzed (Participants) | 39 | 44
  Anti-FHA [pre-booster] | 19.3 [14.8 to 25.2] | 29.6 [21.5 to 40.7]
  Anti-FHA [post-booster]: number analyzed (Participants) | 52 | 54
  Anti-FHA [post-booster] | 358.3 [290.5 to 442.0] | 484.3 [418.9 to 559.9]
  Anti-PRN [pre-booster]: number analyzed (Participants) | 41 | 45
  Anti-PRN [pre-booster] | 15.0 [10.7 to 20.9] | 15.4 [11.3 to 21.0]
  Anti-PRN [post-booster] | 314.3 [229.6 to 430.2] | 509.5 [387.0 to 670.9]

19. Secondary Outcome: Concentrations of Antibodies Against Polyribosyl-ribitol Phosphate (PRP).
Description: as for outcome 12
Time Frame: Before and one month after booster vaccination (at Month 0 and Month 1)
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 53 | 55
µg/mL
  Anti-PRP [pre-booster]: number analyzed (Participants) | 51 | 55
  Anti-PRP [pre-booster] | 0.66 [0.48 to 0.90] | 0.84 [0.64 to 1.12]
  Anti-PRP [post-booster] | 58.26 [43.71 to 77.66] | 49.36 [37.40 to 65.15]

20. Secondary Outcome: Titers of Antibodies Against Poliovirus Types 1, 2 and 3.
Description: Titers were expresses as geometric mean titers (GMTs). The cut-off of the assay was 8.
Time Frame: Before and one month after booster vaccination (at Month 0 and Month 1)
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Number analyzed (Participants) | 28 | 27
Titers
  Anti-polio 1 [pre-booster]: number analyzed (Participants) | 28 | 25
  Anti-polio 1 [pre-booster] | 44.2 [25.3 to 77.1] | 32.8 [19.1 to 56.3]
  Anti-polio 1 [post-booster]: number analyzed (Participants) | 25 | 27
  Anti-polio 1 [post-booster] | 982.2 [688.0 to 1402.3] | 985.2 [627.9 to 1546.0]
  Anti-polio 2 [pre-booster]: number analyzed (Participants) | 28 | 25
  Anti-polio 2 [pre-booster] | 38.0 [25.7 to 56.4] | 34.9 [18.8 to 64.7]
  Anti-polio 2 [post-booster]: number analyzed (Participants) | 25 | 27
  Anti-polio 2 [post-booster] | 1144.1 [773.7 to 1691.7] | 823.4 [553.5 to 1224.8]
  Anti-polio 3 [pre-booster]: number analyzed (Participants) | 28 | 25
  Anti-polio 3 [pre-booster] | 41.0 [24.2 to 69.7] | 43.3 [24.0 to 78.0]
  Anti-polio 3 [post-booster]: number analyzed (Participants) | 25 | 26
  Anti-polio 3 [post-booster] | 1350.8 [857.4 to 2128.2] | 1527.4 [1016.6 to 2294.7]

ADVERSE EVENTS:
Time Frame: Solicited AEs: Within 4 days (Days 0-3) after booster vaccination. SAEs: During the entire study period, from the booster vaccination, at Month 0, up to the study end, at Month 1. Unsolicited AEs:Within 31 days (Days 0-30) after booster vaccination.
Description: Systematically assessed Other Adverse Events are reported only for those participants who completed their symptoms sheet.
Arm/Group | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group
Serious Adverse Events (participants affected / at risk) | 0/118 | 4/120
Other Adverse Events (participants affected / at risk) | 98/118 | 108/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group (N=118) | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group (N=120)
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Bronchiolitis (Infections and infestations) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Synflorix™ Clinical-Commercial + Infanrix™-IPV/Hib Group (N=118) | Synflorix™ Commercial-Commercial + Infanrix™-IPV/Hib Group (N=120)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 6
Pain (General disorders) | 61/117 | 70/117
Redness (General disorders) | 66/117 | 61/117
Swelling (General disorders) | 45/117 | 49/117
Drowsiness (General disorders) | 38/117 | 49/117
Fever (General disorders) | 56/117 | 75/117
Irritability (General disorders) | 51/117 | 67/117
Loss of appetite (General disorders) | 42/117 | 49/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.